CLINICAL TRIAL: NCT00085891
Title: A 6-Week, Multicenter, Double-Blind, Double-Dummy, Randomized Comparison of the Efficacy and Safety of Sustained-Release Formulation Quetiapine Fumarate (SEROQUEL) and Placebo in the Treatment of Acutely Ill Patients With Schizophrenia
Brief Title: Efficacy & Safety of Quetiapine Fumarate (SEROQUEL) & Placebo in the Treatment of Acutely Ill Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1444C00133
Record Dates: First submitted 2004-06-16; First posted 2004-06-18 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenic disorder
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate

SUMMARY:
The purpose of this study is to demonstrate superior efficacy of sustained release quetiapine compared to placebo in patients with schizophrenia after receiving treatment for up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide written informed consent before beginning any study related procedures
* Patient has a documented clinical diagnosis of schizophrenia
* Patient is able to understand and comply with the requirements of the study, as judged by a study investigator

Exclusion Criteria:

* Patients with a history of non-compliance as judged by the study investigator
* Patients with a known lack of response to previous treatment with quetiapine
* Patients who have participated in another drug study within 4 weeks prior to enrollment into this study
* Patients who have previously participated in this study or study D1444C00132

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535
Dates: Start 2004-06; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the Positive and Negative Syndrome Scale (PANSS) total score at the end of treatment.

SECONDARY OUTCOMES:
Evaluation of secondary PANSS efficacy variables and Clinical Global Impression (CGI) variables at all study visits compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (29):
- United States (29):
  - Research Site, Birmingham, Alabama
  - Research Site, Cerritos, California
  - Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Miami, Florida
  - Oak Brook, Illinois
  - Research Site, Oakbrook Terrace, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Rockville, Maryland
  - Brighton, Massachusetts
  - Research Site, Jackson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Holliswood, New York
  - Research Site, Lawrence, New York
  - Research Site, Staten Island, New York
  - Research Site, Medina, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Norristown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Kirkland, Washington